CLINICAL TRIAL: NCT01170871
Title: Phase I Clinical Trial of Ixabepilone and Pemetrexed in Advanced Solid Tumors
Brief Title: Ixabepilone and Pemetrexed/Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor withdrew support
Sponsor: University of Southern California (Other)
Responsible Party: Agustin Garcia, MD, University of Southern California
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0C-08-2
Record Dates: First submitted 2009-11-04; First posted 2010-07-27 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — ixabepilone; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): Escalating doses of Ixabepilone and Pemetrexed
  Interventions: Drug: Ixabepilone; Drug: Pemetrexed

INTERVENTIONS:
Drug: Ixabepilone
Drug: Pemetrexed

SUMMARY:
The purpose of the study is to determine the maximal tolerated dose (MTD) of Ixabepilone and Pemetrexed in advanced solid tumors and to obtain preliminary information regarding the activity of this combination.

This research study is for research participants who have confirmed metastatic or unresectable solid tumors (lung, breast, ovary, cervix, uterus, mesothelioma, and prostate) for which standard curative or palliative measures do not exist or no longer effective.

ELIGIBILITY:
Inclusion Criteria:

* SWOG performance status of 0-2.
* Projected life expectancy of at least 3 months.
* Female and or male age 18 years and over.
* Provision of informed consent prior to any study-related procedures.
* Female patients must not be pregnant due to the potential mutagenicity. and teratogenicity of this treatment. A pregnancy test must be administered 7 days prior to administration of therapy to women of childbearing potential.
* Negative pregnancy test for women of childbearing potential.
* Patients must agree to use some form of contraception while on this study at initiation and for the duration of participation in the study. Sexually active males must also use a reliable and appropriate method of contraception. Post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
* Patients must have recovered from acute toxicities from previous surgery, chemotherapy or radiation therapy.
* Adequate organ function defined as:

  * ANC > 1500/mm3
  * Platelet count > 100,000 cells/mm3
  * Hemoglobin > 9.0g/dL
  * Serum creatinine < 1.5 mg/dl or creatinine clearance > 45 mL/minute
  * (calculated by Cockcroft-Gault formula.)
  * Hepatic function: Patients must have adequate liver functions: AST or ALT < 2.5 X upper limit of normal (ULN), alkaline phosphatase < 2.5 X upper limit of normal. In patients with bone metastasis and no evidence of liver metastasis and bilirubin < upper limit of normal an alkaline phosphatase < 5 ULN will be allowed
  * Serum Bilirubin < 1.5 mg/dL
* Peripheral neuropathy grade 0-1.
* No other concomitant therapy directed at the cancer is allowed.
* The ability to interrupt NSAIDS 2 days before (5 days for long-acting NSAIDs), the day of, and 2 days following administration of pemetrexed.
* The ability to take folic acid, Vitamin B12, and dexamethasone according to protocol.

Exclusion Criteria:

* Laboratory results:

  * Serum bilirubin > 1.5 the upper limit of reference range (ULRR)
  * Serum creatinine >1.5 x ULRR or creatinine clearance < 45 mL/minute (calculated by Cockcroft-Gault formula)
* Women who are currently pregnant or breast feeding.
* Receipt of any investigational agents within 30 days prior to commencing study treatment.
* Last dose of prior chemotherapy discontinued less than 4 weeks before the start of study therapy.
* Last radiation therapy within the last 4 weeks before the start of study therapy, except palliative radiotherapy.
* Prior radiation must not have included ≥ 30% of major bone marrow containing areas (pelvis, lumbar spine).
* Any unresolved toxicity greater than CTC grade 1 from previous anti- cancer therapy, excluding alopecia.
* CTC Grade 1 or greater neuropathy (motor or sensory) at study entry.
* Hematologic function with absolute neutrophils ≤ 1500/mm3 and/or platelets < 100,000/mm 3.
* Hepatic function with serum bilirubin greater than the upper institutional limits of normal, ALT and AST > 2.5 times the upper institutional limits of normal.
* Presence of third space fluid which cannot be controlled by drainage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
To determine the maximal tolerated dose (MTD) of Ixabepilone and Pemetrexed in advanced solid tumors. | weekly

SECONDARY OUTCOMES:
Response Rate | every 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Agustin Garcia, MD, Principal Investigator — Univrsity of Southern California
Locations (2):
- United States (2):
  - Los Angeles County+University of Southern California Medical Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California